CLINICAL TRIAL: NCT00481650
Title: A Prospective Observation Study (Anwendungsbeobachtung [AWB]) of the Prescribing and Administration Practices of German Gynecologists With Leios® Dragées/Alesse
Brief Title: Observational Trial With Leios/Alesse
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 101742
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Contraceptives, Oral, Combined
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Leios/Alesse

SUMMARY:
A prospective, observational study (Anwendungsbeobachtung [AWB]) of the prescribing and administration practices of German gynecologists with Leios® Dragées.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, women, aged under 40

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 2005-05; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com